CLINICAL TRIAL: NCT03608423
Title: The Dutch Intracerebral Hemorrhage Surgery Trial Pilot Study; Minimally-invasive Endoscopy-guided Surgery for Spontaneous Intracerebral Hemorrhage
Brief Title: Dutch Intracerebral Hemorrhage Surgery Trial Pilot Study
Acronym: DIST pilot
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: Dutch Heart Foundation (Other); Penumbra Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NL6310007817
Record Dates: First submitted 2018-04-30; First posted 2018-08-01 (Actual); Last update posted 2022-10-13 (Actual); Status verified 2022-08

CONDITIONS: Intracerebral Hemorrhage; Surgical Procedures, Minimally Invasive
Keywords: Intracerebral Hemorrhage; Surgical Procedures, Minimally Invasive; Surgical Procedures, Endoscopic
MeSH Terms: conditions — Cerebral Hemorrhage

STUDY DESIGN:
Intervention Model Description: We will include 40 patients in the surgical arm (inclusion in three hospitals) and aim for 120 matched controls in the other arm (in 7 other hospitals).
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Surgical treatment (Experimental): Minimally-invasive endoscopy-guided surgery or hematoma aspiration, additional to standard medical treatment.
  Interventions: Device: Minimally-invasive endoscopy-guided surgery
- Standard medical management (No Intervention): Standard medical treatment (treatment of bloodpressure, admission to stroke unit and supportive care, surgical treatment if necessary in case of deterioration)

INTERVENTIONS:
Device: Minimally-invasive endoscopy-guided surgery — Surgery started within 8 hours of onset of spontaneous intracerebral hemorrhage.
  Other Names: Minimally-invasive endoscopy-guided hematoma aspiration
  Arms: Surgical treatment

SUMMARY:
Background:

Intracerebral hemorrhage (ICH) accounts for 15-20% of all strokes in Western Europe, and contributes profoundly to mortality and disability. Thirty day case fatality is 40% and of those surviving, only few gain independence. Except for stroke unit care and early blood pressure lowering there is currently no treatment of proven benefit. Important predictors of poor outcome are increasing age, decreasing Glasgow Coma Scale score, increasing ICH volume, presence of intraventricular hemorrhage and deep or infratentorial location. In addition, secondary injury due to development of edema and inflammatory response, contribute to disability and death. Surgical treatment, mostly comprising craniotomy, has so far not been proven effective. In the largest trials STICH and STICH II, the median time to treatment was more than 24 hours, which may be an important explanation for the lack of treatment effect.

The investigators hypothesize that early, minimally-invasive, endoscopy-guided surgery improves outcome in patients with spontaneous supratentorial ICH.

Objective: to study safety, feasibility and technical effectiveness of minimally-invasive endoscopy guided surgery for treatment of spontaneous supratentorial ICH and to estimate the potential effect on outcome.

Study design: a multicenter, prospective intervention study (phase II) with a telephonic follow up interview at 90 and 180 days.The pilot study serves as a prelude to a randomized phase III trial in which the investigators aim to assess whether this intervention improves functional outcome at 90 and 180 days.

Study population: patients with spontaneous supratentorial ICH of 18 years and older. Forty patients in three participating centers (Radboudumc, Erasmus MC and AMC) will undergo minimally-invasive endoscopy-guided surgery. Three-hundred-and-sixty patients undergoing standard medical treatment in one of 7 other participating centers, will be included as a control group.

Intervention: minimally-invasive endoscopy-guided surgery within 8 hours of symptom onset, in addition to standard medical management.

Primary study outcomes: safety (death within 24 hours, 7-day procedure related complications, 7-day mortality, 30-day mortality) and technical effectiveness (proportional volume reduction, proportion of participants with volume reduction > 60 and >80%, and proportion with remaining clot volume <15mL).

Secondary outcomes: modified Rankin Scale score at 90 and 180 days after ICH (functional outcome).

DETAILED DESCRIPTION:
The full protocol is available at https://dutch-ich.nl/trial-protocol-and-trial-documents.html

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18
2. NIHSS ≥ 2
3. Supratentorial ICH confirmed by CT, without a CT-angiography confirmed causative vascular lesion (e.g. aneurysma, arteriovenous malformation [AVM], dural arteriovenous fistula [DAVF], cerebral venous sinus thrombosis [CVST]).
4. Minimal lesion size 10 mL
5. Intervention can be started within 8 hours from symptoms onset; or for controls presentation within 8 hours of symptom onset.
6. Patient's or legal representative's written informed consent

Exclusion Criteria:

1. Pre-stroke disability, which interferes with the assessment of functional outcome at 90 days, i.e. mRS > 2
2. Causative vascular lesion (e.g. aneurysm, AVM, DAVF, CVST) on CT-angiography or other known underlying cause (e.g. tumor, cavernoma)
3. Untreated coagulation abnormalities, including INR > 1.3 (point of care measurement allowed) and treatment with oral thrombin or factor X antagonists; patients on vitamin K antagonist can be included after correction of the INR.
4. Current known severe infection for which antibiotic treatment at time of ICH symptom onset
5. Patient moribund (e.g. coning, bilateral dilated unresponsive pupils)
6. Pregnancy (note: most patients will be beyond child bearing age; if not a pregnancy test is mandatory).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 169 (Actual)
Dates: Start 2018-12-03 (Actual); Primary Completion 2022-04-07 (Actual); Study Completion 2022-04-07 (Actual)

PRIMARY OUTCOMES:
Death within 24 hours | 24 hours
  Death within 24 hours after baseline.
Neurological deterioration within 24 hours | 24 hours
  Neurological deterioration, defined as an increase of ≥4 points on the sumscore of the NIHSS or >2 National Institutes of Health Stroke Scale (NIHSS)is a sum score, composed of 11 items, each of which scores a specific ability between 0 and 4. For each item, a score of 0 typically indicates normal function in that ability, while a higher score indicates the level of impairment. The total score varies between 0 (no symptoms at all) and 42. points on one item of NIHSS,
Proportion of volume reduction | Baseline and 24 hours (based on the comparison baseline CT and CT at 24 hours).
  The proportion of volume reduction, based on baseline CT and CT at 24 hours (in the intervention group).

SECONDARY OUTCOMES:
Procedure related complications | 7 days
  The proportion of patients with procedure related complications at 7 days, including: rebleed, intracranial hemorrhage, epileptic seizures and intracranial infection. (in the intervention group)
Mortality at 7 days | 7 days
  Proportion of patients that died within 7 days after baseline
Mortality at 30 days | 30 days
  Proportion of patients that died within 30 days after baseline
Percentage of patients with clot volume reduction ≥60% | Baseline and 24 hours CT (the difference is measured)
  The proportion of patients in which the clot volume could be reduced with 60% or more, based on the comparison baseline CT and CT at 24 hours. (in the intervention group)
Percentage of patients with clot volume reduction ≥ 80% | Baseline and 24 hours CT (the difference is measured)
  The proportion of patients in which the clot volume could be reduced with 80% or more, based on the comparison baseline CT and CT at 24 hours. (in the intervention group)
Percentage of patients with remaining clot volume of ≤ 15mL | 24 hours CT
  The proportion of patients in which due to clot removal a remaining clot volume of ≤ 15mL was established at 24 hours. (in the intervention group)
Proportion of conversion to craniotomy | 24 hours
  The proportion of patients in which a conversion to craniotomy was required and done. (in the intervention group)
Functional outcome at 3 months | 3 months (90 days)
  Ordinal shift in functional outcome (comparing the intervention group to the controls), assessed with the modified Rankin Scale (mRS) at 3 months. This is a six point scale in which a score of 0 means no symptoms at all, a higher score means more impairment, and a score of 6 means the participant is dead.
  A favorable outcome is defined as mRS 0-3 and mRS 0-2.
Functional outcome at 6 months | 6 months (180 days)
  Ordinal shift in functional outcome (comparing the intervention group to the controls), , assessed with the modified Rankin Scale (mRS) at 6 months. This is a six point scale in which a score of 0 means no symptoms at all, a higher score means more impairment, and a score of 6 means the participant is dead.
  A favorable outcome is defined as mRS 0-3 and mRS 0-2.
National Institute of Health Stroke Scale (NIHSS) at 7 days or discharge | 7 days (or at discharge from the hospital if earlier)
  National Institutes of Health Stroke Scale (NIHSS)is a sum score, composed of 11 items, each of which scores a specific ability between 0 and 4. For each item, a score of 0 typically indicates normal function in that ability, while a higher score indicates the level of impairment. The total score varies between 0 (no symptoms at all) and 42.

CONTACTS AND LOCATIONS:
Overall Officials: Ruben Dammers, Dr., Principal Investigator — Erasmus Medical Center
Locations (10):
- Netherlands (10):
  - Radboud University Medical Center, Nijmegen, Gelderland
  - Academic Medical Center, Amsterdam
  - Medisch Spectrum Twente, Enschede
  - Leiden University Medical Center, Leiden
  - Maastricht University Medical Center, Maastricht
  - Erasmus Medical Center, Rotterdam
  - Haaglanden Medical Center, The Hague
  - Elisabeth Tweesteden Ziekenhuis, Tilburg
  - University Medical Center Utrecht, Utrecht
  - Isala, Zwolle

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Sondag L, Schreuder FHBM, Pegge SAH, Coutinho JM, Dippel DWJ, Janssen PM, Vandertop WP, Boogaarts HD, Dammers R, Klijn CJM; Dutch ICH Surgery Trial Study Group, part of the CONTRAST consortium. Safety and technical efficacy of early minimally invasive endoscopy-guided surgery for intracerebral haemorrhage: the Dutch Intracerebral haemorrhage Surgery Trial pilot study. Acta Neurochir (Wien). 2023 Jun;165(6):1585-1596. doi: 10.1007/s00701-023-05599-2. Epub 2023 Apr 27. PMID 37103585
- [Derived] Lahr MMH, Maas WJ, van der Zee DJ, Uyttenboogaart M, Buskens E. Rationale and design for studying organisation of care for intra-arterial thrombectomy in the Netherlands: simulation modelling study. BMJ Open. 2020 Jan 7;10(1):e032754. doi: 10.1136/bmjopen-2019-032754. PMID 31915166
- See also: Website of the Dutch ICH Surgery Trial pilot study — http://dutch-ich.nl